CLINICAL TRIAL: NCT05922631
Title: Effect of Airway Pressure Release Ventilation vs. Low Tidal Volume Ventilation on Right Heart Function in Acute Respiratory Distress Syndrome Patients: a Single-center Randomized Controlled Study
Brief Title: Effect of APRV vs. LTV on Right Heart Function in ARDS Patients: a Single-center Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: XiaoJing Zou,MD (Other)
Responsible Party: Sponsor-Investigator, XiaoJing Zou,MD, Clinical Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALRVD2022
Record Dates: First submitted 2023-06-19; First posted 2023-06-28 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-05

CONDITIONS: Right Heart Failure; Mechanical Ventilation; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Heart Failure; Respiratory Distress Syndrome | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Patients with ARDS who met the inclusion criteria were randomized to APRV or LTV mechanical ventilation. Ventilator parameters were set according to the study protocol, P high: Tidal volume (VT) was set at 6ml/kg of ideal body weight, and plateau pressure (Pplat) was measured. Initial Phigh was set at Pplat, usually 20-32 cmH2O. The APRV end-expiratory flow rate was set at 75% of the peak expiratory flow rate. For LTV mechanical ventilation, ARDSnet method was used to set the tidal volume according to 4-8ml/kg, so that Pplat<30cmH2O
Who Masked: Participant
Masking Description: participants are blinded to accept APRV or LTV after inclusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- APRV group (Experimental): In APRV group, ventilator parameters were set according to the study protocol, P high: Tidal volume (VT) was set at 6ml/kg of ideal body weight, and plateau pressure (Pplat) was measured. Initial Phigh was set at Pplat, usually 20-32 cmH2O. The APRV end-expiratory flow rate was set at 75% of the peak expiratory flow rate.
  Interventions: Procedure: Airway pressure release ventilation
- LTV group (Placebo Comparator): The ARDSnet method was used for LTV group mechanical ventilation, and the tidal volume was set according to 4-8ml/kg, so that the Pplat was <30cmH2O
  Interventions: Procedure: low tidal volume

INTERVENTIONS:
Procedure: Airway pressure release ventilation — ventilator parameters were set according to the study protocol, P high: Tidal volume (VT) was set at 6ml/kg of ideal body weight, and plateau pressure (Pplat) was measured. Initial Phigh was set at Pplat, usually 20-32 cmH2O. The APRV end-expiratory flow rate was set at 75% of the peak expiratory flow rate.
  Arms: APRV group
Procedure: low tidal volume — The ARDSnet method was used for LTV mechanical ventilation, and the tidal volume was set according to 4-8ml/kg, so that the Pplat was <30cmH2O
  Arms: LTV group

SUMMARY:
Acute Respiratory Distress Syndrome (ARDS) is often complicated by Right Ventricular Dysfunction (RVD), and the incidence can be as high as 64%. The mechanism includes pulmonary vascular dysfunction and right heart systolic dysfunction. Pulmonary vascular dysfunction includes acute vascular inflammation, pulmonary vascular edema, thrombosis and pulmonary vascular remodeling. Alveolar collapse and over distension can also lead to increased pulmonary vascular resistance, Preventing the development of acute cor pulmonale in patients with acute respiratory distress. ARDS patients with RVD have a worse prognosis and a significantly increased risk of death, which is an independent risk factor for death in ARDS patients. Therefore, implementing a right heart-protective mechanical ventilation strategy may reduce the incidence of RVD.

APRV is an inverse mechanical ventilation mode with transient pressure release under continuous positive airway pressure, which can effectively improve oxygenation and reduce ventilator-associated lung injury. However, its effect on right ventricular function is still controversial. Low tidal volume (LTV) is a mechanical ventilation strategy widely used in ARDS patients. Meta-analysis results showed that compared with LTV, APRV improved oxygenation more significantly, reduced the time of mechanical ventilation, and even had a tendency to improve the mortality of ARDS patients However, randomized controlled studies have shown that compared with LTV, APRV improves oxygenation more significantly and also increases the mean airway pressure. Therefore, some scholars speculate that APRV may increase the intrathoracic pressure, pulmonary circulatory resistance, and the risk of right heart dysfunction but this speculation is not supported by clinical research evidence. In addition, APRV may improve right ventricular function by correcting hypoxia and hypercapnia, promoting lung recruitment and reducing pulmonary circulation resistance. Therefore, it is very important to clarify this effect for whether APRV can be safely used and popularized in clinic.we aim to conduct a single-center randomized controlled study to further compare the effects of APRV and LTV on right ventricular function in patients with ARDS, pulmonary circulatory resistance (PVR) right ventricular-pulmonary artery coupling (RV-PA coupling), and pulmonary vascular resistance (PVR).

DETAILED DESCRIPTION:
Acute Respiratory DistressSyndrome (ARDS) is often complicated by Right Ventricular Dysfunction (RVD), and the incidence can be as high as 64%. The mechanism includes pulmonary vascular dysfunction and right heart systolic dysfunction. Pulmonary vascular dysfunction includes acute vascular inflammation, pulmonary vascular edema, thrombosis and pulmonary vascular remodeling. Alveolar collapse and alveolar overdistension can also lead to increased pulmonary vascular resistance, Preventing the development of acute cor pulmonale in patients with acute respiratory distress. ARDS patients with RVD have a worse prognosis and a significantly increased risk of death, which is an independent risk factor for death in ARDS patients [2-4]. Therefore, implementing a right heart-protective mechanical ventilation strategy may reduce the incidence of RVD.

Mechanical ventilation is the main treatment for moderate to severe ARDS. Mechanical ventilation promotes lung recruitment and reduces mechanical compression of pulmonary vessels between alveoli and alveolar walls. In addition, mechanical ventilation corrected hypoxemia and hypercapnia, thereby reducing reactive pulmonary vasoconstriction. All of the above can reduce pulmonary circulation resistance and right ventricular afterload, thereby improving right ventricular function in patients with ARDS. However, if hyperventilation occurs, it will increase the mechanical compression of pulmonary vessels on the alveolar wall, increase the intrathoracic pressure, and increase the afterload of the right heart, which will adversely affect the function of the right heart. There are a variety of ventilation strategies for patients with ARDS in clinical practice, but which mechanical ventilation has the protective function of right heart or has little effect on right heart function, so far there is a lack of relevant research reports.

Airway pressure release ventilation (APRV) is an inverse mechanical ventilation mode with transient pressure release under continuous positive airway pressure, which can effectively improve oxygenation and reduce ventilator-associated lung injury. However, its effect on right ventricular function is still controversial, so its clinical application is not popular, and it is only used as one of the salvage treatments for ARDS patients. Low tidal volume (LTV) is a mechanical ventilation strategy widely used in ARDS patients, but it does not further reduce mortality in patients with moderate to severe ARDS. Meta-analysis results showed that compared with LTV, APRV improved oxygenation more significantly, reduced the time of mechanical ventilation, and even had a tendency to improve the mortality of ARDS patients [7]. However, randomized controlled studies have shown that compared with LTV, APRV improves oxygenation more significantly and also increases the mean airway pressure [8]. Therefore, some scholars speculate that APRV may increase the intrathoracic pressure, pulmonary circulatory resistance, and the risk of right heart dysfunction , but this speculation is not supported by clinical research evidence. In addition, the results of animal experiments suggest that APRV improves oxygenation, promotes lung recruitment, and improves the heterogeneity of lung lesions in ARDS, without causing lung hyperventilation, suggesting that APRV may not increase pulmonary circulatory resistance. In addition, APRV may improve right ventricular function by correcting hypoxia and hypercapnia, promoting lung recruitment and reducing pulmonary circulation resistance. Therefore, the impact of APRV on right ventricular function is still unclear, and it is very important to clarify this effect for whether APRV can be safely used and popularized in clinic. Therefore, our research group conducted a prospective observational study, "The effect of APRV on right ventricular function evaluated by Transthoracic Echocardiography, [2022] Lun Lun Zi (0075)". The study results suggested that APRV improved lung perfusion in ARDS patients while effectively improving oxygenation and promoting lung recruitment. The incidence of RVD was not increased, and there was no hemodynamic deterioration in ARDS patients. APRV is safe and effective for patients with ARDS. However, the results of a single-arm prospective observational study with a small sample size cannot provide strong evidence for clinical practice. In the previous studies, all the right ventricular function was assessed by transthoracic echocardiography. Due to the limitation of the sound window of transthoracic echocardiography, the right ventricular function of some ARDS patients could not be evaluated. Therefore, this study intends to use transesophageal echocardiography or transthoracic echocardiography to fully evaluate the right ventricular function of all enrolled patients as much as possible, and to conduct a single-center randomized controlled study to further compare the effects of APRV and LTV on right ventricular function in patients with ARDS, pulmonary circulatory resistance (PVR), right ventricular-pulmonary artery coupling (RV-PA coupling), and pulmonary vascular resistance (PVR).Whether there are different effects on hemodynamics and mortality. It is hoped that the results of this study will provide more evidence support for the clinical application of APRV and benefit more ARDS patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients who meet the 2012 Berlin ARDS diagnostic criteria and perform invasive mechanical ventilation 2, PEEP≥5cmH2O, oxygenation index ≤200mmHg 3. Tracheal intubation and mechanical ventilation were performed for less than 48h at the time of inclusion 4. Age ≥18 years and ≤80 years

Exclusion Criteria:

* 1.abdominal pressure≥20mmHg 2.BMI≥35kg/m2; 3. pregnant and lactating women 4.expected duration of invasive mechanical ventilation < 72 hours 5. neuromuscular diseases known to require prolonged mechanical ventilation 6.severe chronic obstructive pulmonary disease, severe asthma, Interstitial lung disease 7.intracranial hypertension, 8.pulmonary bullae or pneumothorax, subcutaneous emphysema, or mediastinal emphysema, 9.extracorporeal membrane oxygenation or prone position ventilation on admission to the ICU 10. uncorrected shock of various types and refractory shock 11.pulmonary embolism 12.severe cardiac dysfunction (New York Heart Association class III or IV). Acute coronary syndrome or sustained ventricular tachyarrhythmia), right heart enlargement due to chronic cardiopulmonary diseases, cardiogenic shock or after major cardiac surgery 13.poor cardiac sound window, unable to obtain cardiac ultrasound images 14.no informed consent was signed

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence of right heart dysfunction in ARDS patients with APRV or LTV mechanical ventilation for 24h | at the time of 24 hours after inclusion
  Incidence of right heart dysfunction in ARDS patients with APRV or LTV mechanical ventilation for 24h.Abnormal findings on any of the following ultrasound measures can be considered as right ventricular dysfunction, including: tricuspid annular plane systolic excursion (TAPSE) <17 mm, tricuspid annular plane systolic velocity (S') <9.5 cm/s, right ventricular fractional area change (FAC) <35%, ratio of right ventricular end-diastolic area to left ventricular end-diastolic area (RVEDA/LVEDA) >0.6, or right ventricular to left ventricular end-diastolic diameter ratio (RV/LV ratio) >1.

SECONDARY OUTCOMES:
Incidence of right heart dysfunction in ARDS patients with APRV or LTV mechanical ventilation for 48h | at the time of 48 hours after inclusion
  Incidence of right heart dysfunction in ARDS patients with APRV or LTV mechanical ventilation for 24h.Abnormal findings on any of the following ultrasound measures can be considered as right ventricular dysfunction, including: right ventricular end-diastolic diameter/left ventricular end-diastolic diameter(RVEDD/LVEDD)>1.0, right ventricular fractional area change(FAC)<35%,tricuspid annular plane systolic excursion(TAPSE)<17mm,Systolic S'velocity of tricuspid annulus <9.5 cm/s by TDI
Incidence of right heart dysfunction in ARDS patients with APRV or LTV mechanical ventilation for 72h | at the time of 72 hours after inclusion
  Incidence of right heart dysfunction in ARDS patients with APRV or LTV mechanical ventilation for 24h.Abnormal findings on any of the following ultrasound measures can be considered as right ventricular dysfunction, including: right ventricular end-diastolic diameter/left ventricular end-diastolic diameter(RVEDD/LVEDD)>1.0, right ventricular fractional area change(FAC)<35%,tricuspid annular plane systolic excursion(TAPSE)<17mm,Systolic S'velocity of tricuspid annulus <9.5 cm/s by TDI
Values of tricuspid annular plane systolic excursion at 24th hour | at the time of 24 hours after inclusion
  Tricuspid annular plane systolic excursion(TAPSE) was measured by echocardiography in the apical four-chamber view, using M mode measurements, with the sampling line aligned to the tricuspid annulus.
Values of tricuspid annular plane systolic excursion at 48th hour | at the time of 48 hours after inclusion
  Tricuspid annular plane systolic excursion(TAPSE) was measured by echocardiography in the apical four-chamber view, using M mode measurements, with the sampling line aligned to the tricuspid annulus.
Values of tricuspid annular plane systolic excursion at 72th hour | at the time of 72 hours after inclusion
  Tricuspid annular plane systolic excursion(TAPSE) was measured by echocardiography in the apical four-chamber view, using M mode measurements, with the sampling line aligned to the tricuspid annulus.
Values of right ventricular end-diastolic diameter/left ventricular end-diastolic diameter(RVEDD/LVEDD) at 24th hour | at the time of 24 hours after inclusion
  The maximum transverse diameter of the right/left ventricular inflow tract near the basal 1/3 was measured in the apical four-chamber view
Values of right ventricular end-diastolic diameter/left ventricular end-diastolic diameter(RVEDD/LVEDD) at 48th hour | at the time of 48 hours after inclusion
  The maximum transverse diameter of the right/left ventricular inflow tract near the basal 1/3 was measured in the apical four-chamber view
Values of right ventricular end-diastolic diameter/left ventricular end-diastolic diameter(RVEDD/LVEDD) at 72th hour | at the time of 72 hours after inclusion
  The maximum transverse diameter of the right/left ventricular inflow tract near the basal 1/3 was measured in the apical four-chamber view
Values of right ventricular fractional area change(RVFAC) at 24th hour | at the time of 24 hours after inclusion
  RVFAC = (end-diastolic area - end-systolic area)/end-diastolic area ×100%.The right ventricle is shown in the apical four-chamber cardiac view.
Values of right ventricular fractional area change(RVFAC) at 48th hour | at the time of 48 hours after inclusion
  RVFAC = (end-diastolic area - end-systolic area)/end-diastolic area ×100%.The right ventricle is shown in the apical four-chamber cardiac view.
Values of right ventricular fractional area change(RVFAC) at 72th hour | at the time of 72 hours after inclusion
  RVFAC = (end-diastolic area - end-systolic area)/end-diastolic area ×100%.The right ventricle is shown in the apical four-chamber cardiac view.
Values of Systolic S'velocity of tricuspid annulus by at 24th, 48th and 72th hour | at the time of 24 hours (h), 48h and 72h after inclusion
  Tissue Doppler sampling volume is placed in the middle of the right ventricular tricuspid annulus or basal segment of the right ventricular free wall to measure systolic velocity S'.
Values of hemodynamic measures at 24th, 48th and 72th hour | at the time of 24 hours (h), 48h and 72h after inclusion
  hemodynamic measures including: heart rate, mean arterial pressure,central venous pressure,Dose of vasoactive agents accumulated over 24 hours,cumulative fluid balance over 24 hours.
Values of respiratory mechanics parameters at 24th, 48th and 72th hour | at the time of 24 hours (h), 48h and 72h after inclusion
  Respiratory mechanics parameters including Peak pressure, Plateau pressure,Driving pressure,Respiratory system compliance and Airway resistance are measured by using routine procedures
28-day mortality | Day 28 after study entry
  28-day mortality after study entry
in hospital mortality | Maximum 90-day in-hospital mortality
  in hospital mortality after study entry
28 days of ventilator free days | Day 28 after study entry
  28 days of ventilator free days after study entry
Values of arterial partial pressure of oxygen/fraction of inspired oxygen at 24th, 48th and 72th hour | at the time of 24 hours (h), 48h and 72h after inclusion
  arterial partial pressure of oxygen/fraction of inspired oxygen are measured at 24th, 48th and 72th hour after inclusion
Values of arterial partial pressure of carbon dioxide at 24th, 48th and 72th hour | at the time of 24 hours (h), 48h and 72h after inclusion
  arterial partial pressure of carbon dioxide are measured at 24th, 48th and 72th hour after inclusion
ventilation ratio at 24th, 48th and 72th hour | at the time of 24 hours (h), 48h and 72h after inclusion
  VR=[minute ventilation ×PaCO2]/[predicted body weight ×100×37.5]
Incidence prone position ventilation during hospitalization | Day 28 after study entry
  Incidence of prone position ventilation during hospitalization after study entry
ventilator settings at 24th, 48th and 72th hour | at the time of 24 hours (h), 48h and 72h after inclusion
  ventilator settings including minute ventilation, Fraction of inspired oxygen, tidal volume, positive end-expiratory pressure, respiratory rate, mean airway pressure
Velocity-time integral of left ventricular outflow tract at 24th, 48th and 72th hour | at the time of 24 hours (h), 48h and 72h after inclusion
  Velocity-time integral(Vti) of left ventricular outflow tract are measured at the apical five-chamber heart view. The sampling volume was placed in the left ventricular outflow tract, below the aortic valve, in pulsed Doppler mode with a window width of 2-4mm. The velocity time integral (VTI) image of aortic blood flow can be obtained by placing the sampling volume below the aortic valve orifice , adjusting the probe so that the direction of blood flow is as parallel as possible to the sampling line, and selecting the pulsed Doppler mode (PW)
Stroke volume at 24th, 48th and 72th hour | at the time of 24 hours (h), 48h and 72h after inclusion
  Stroke volume(SV)=15.VTI×π(D/2)*(D/2), D=Left ventricular outflow tract diameter(LVOT diameter)
cardiac output at 24th, 48th and 72th hour | at the time of 24 hours (h), 48h and 72h after inclusion
  cardiac output(CO)=SV*HR
Velocity-time integral of right ventricular outflow tract at 24th, 48th and 72th hour | at the time of 24 hours (h), 48h and 72h after inclusion
  Velocity-time integral(Vti) of right ventricular outflow tract are measured at the view of the right ventricular outflow tract. The sampling volume was placed in the right ventricular outflow tract, below the aortic valve, in pulsed Doppler mode with a window width of 2-4mm. The velocity time integral (VTI) image of aortic blood flow can be obtained by placing the sampling volume below the aortic valve orifice , adjusting the probe so that the direction of blood flow is as parallel as possible to the sampling line, and selecting the pulsed Doppler mode (PW)
Tricuspid annular diameter | at the time of 24 hours (h), 48h and 72h after inclusion
  Tricuspid annular diameters are measured at the apical four-chamber heart view
The velocity of tricuspid regurgitation | at the time of 24 hours (h), 48h and 72h after inclusion
  The velocity of tricuspid regurgitation are measured at the apical four-chamber heart view.The CW Doppler sampling line was placed at the tricuspid valve orifice.
Length of hospital stay | Maximum 90-day hospital stay
  hospital stay after hospital entry
Length of ICU stay | Maximum 90-day ICU stay
  hospital stay after ICU entry
Incidence of tracheotomy | Day 28 after study entry
  Incidence of tracheotomy during hospitalization after study entry

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojing zou, MD, Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Background] Zhang H, Huang W, Zhang Q, Chen X, Wang X, Liu D; Critical Care Ultrasound Study Group. Prevalence and prognostic value of various types of right ventricular dysfunction in mechanically ventilated septic patients. Ann Intensive Care. 2021 Jul 13;11(1):108. doi: 10.1186/s13613-021-00902-9. PMID 34255224
- [Background] Boissier F, Katsahian S, Razazi K, Thille AW, Roche-Campo F, Leon R, Vivier E, Brochard L, Vieillard-Baron A, Brun-Buisson C, Mekontso Dessap A. Prevalence and prognosis of cor pulmonale during protective ventilation for acute respiratory distress syndrome. Intensive Care Med. 2013 Oct;39(10):1725-33. doi: 10.1007/s00134-013-2941-9. Epub 2013 May 15. PMID 23673401
- [Background] Dong D, Zong Y, Li Z, Wang Y, Jing C. Mortality of right ventricular dysfunction in patients with acute respiratory distress syndrome subjected to lung protective ventilation: A systematic review and meta-analysis. Heart Lung. 2021 Sep-Oct;50(5):730-735. doi: 10.1016/j.hrtlng.2021.04.011. Epub 2021 Jun 9. PMID 34118786
- [Background] Mekontso Dessap A, Boissier F, Charron C, Begot E, Repesse X, Legras A, Brun-Buisson C, Vignon P, Vieillard-Baron A. Acute cor pulmonale during protective ventilation for acute respiratory distress syndrome: prevalence, predictors, and clinical impact. Intensive Care Med. 2016 May;42(5):862-870. doi: 10.1007/s00134-015-4141-2. Epub 2015 Dec 9. PMID 26650055
- [Background] Sipmann FS, Santos A, Tusman G. Heart-lung interactions in acute respiratory distress syndrome: pathophysiology, detection and management strategies. Ann Transl Med. 2018 Jan;6(2):27. doi: 10.21037/atm.2017.12.07. PMID 29430444
- [Background] Cheng J, Ma A, Dong M, Zhou Y, Wang B, Xue Y, Wang P, Yang J, Kang Y. Does airway pressure release ventilation offer new hope for treating acute respiratory distress syndrome? J Intensive Med. 2022 Mar 28;2(4):241-248. doi: 10.1016/j.jointm.2022.02.003. eCollection 2022 Oct. PMID 36785647
- [Background] Sun X, Liu Y, Li N, You D, Zhao Y. The safety and efficacy of airway pressure release ventilation in acute respiratory distress syndrome patients: A PRISMA-compliant systematic review and meta-analysis. Medicine (Baltimore). 2020 Jan;99(1):e18586. doi: 10.1097/MD.0000000000018586. PMID 31895807
- [Background] Zhou Y, Jin X, Lv Y, Wang P, Yang Y, Liang G, Wang B, Kang Y. Early application of airway pressure release ventilation may reduce the duration of mechanical ventilation in acute respiratory distress syndrome. Intensive Care Med. 2017 Nov;43(11):1648-1659. doi: 10.1007/s00134-017-4912-z. Epub 2017 Sep 22. PMID 28936695
- [Background] Andrews P, Shiber J, Madden M, Nieman GF, Camporota L, Habashi NM. Myths and Misconceptions of Airway Pressure Release Ventilation: Getting Past the Noise and on to the Signal. Front Physiol. 2022 Jul 25;13:928562. doi: 10.3389/fphys.2022.928562. eCollection 2022. PMID 35957991
- [Background] Robinson B, Ebeid M. A simple echocardiographic method to estimate pulmonary vascular resistance. Am J Cardiol. 2014 Jan 15;113(2):412. doi: 10.1016/j.amjcard.2013.11.001. Epub 2013 Nov 7. No abstract available. PMID 24387904